CLINICAL TRIAL: NCT06659081
Title: Effect of Subepithelial Connective Tissue Graft with Socket Shield Technique on Periimplant Tissues in Immediate Implant Procedure
Brief Title: Effect of Subepithelial Connective Tissue Graft with Socket Shield Technique
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, osama ahmed mahmoud elnaggar, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-Rec IM122333
Record Dates: First submitted 2024-09-17; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Socket Shield Technique Implant Placement; Immediate Implant Placement
Keywords: partial extraction therapy
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- socket shield technique (Experimental)
  Interventions: Procedure: socket shield technique; Procedure: subepithelial connective tissue graft; Procedure: implant placement
- immediate implant placement (Experimental)
  Interventions: Procedure: subepithelial connective tissue graft; Procedure: implant placement

INTERVENTIONS:
Procedure: socket shield technique — partial extraction therapy : sectioning the root and keeping part of it in contact with labial plate of bone
  Other Names: partial extraction therapy
  Arms: socket shield technique
Procedure: subepithelial connective tissue graft — A connective tissue graft harvesting from maxillary tuberosity area
Procedure: implant placement — implant placement

SUMMARY:
The goal of this clinical trial is to Evaluate of the soft tissue profile changes and labial plate of bone in the anterior esthetic area when using socket shield technique in conjunction with immediate implant and subepithelial connective tissue graft, in comparison to using immediate implant combined by subepithelial connective tissue graft. The main questions it aims to answer is :

* does the socket shield technique better preserve gingival contours and connective tissues, resulting in improved esthetic outcomes?
* Researchers will compare socket shield combined with immediate implant placement and a subepithelial connective tissue graft to immediate implant placement with just a subepithelial connective tissue graft to see if more favorable soft tissue profile changes and better preservation of the labial plate of bone are obtained.

participants will :

. subjected to partially extracted socket with immediately placed implant and subepithelial connective tissue graft.

.subjected to immediate implant with subepithelial connective tissue graft.

ELIGIBILITY:
Inclusion Criteria:

* Medically free
* Maxillary esthetic zone extended to the second premolar with healthy roots
* Good oral hygiene
* Hopeless teeth

Exclusion Criteria:

* Patients with systemic conditions that can affect bone turnover
* Smokers
* Pregnant women
* Chronic and active periodontal disease
* Vertical and horizontal root fracture
* Dehiscence or fenestration of the labial plate of bone
* Gingival recession

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of soft tissue profile around the implant | change from baseline at six months
  - Scanning of preoperative and postoperative cast , then Volumetric analysis of soft tissue by Superimposing the scans to evaluate the changes in the soft tissues in millimeters.

SECONDARY OUTCOMES:
Assessment of labial plate of bone around the implant | change from baseline at six months
  Preoperative CBCT to measure thickness, height and density of existent labial plate of bone in millimeters at baseline. Then, six months later, a CBCT is carried out to measure the difference between these measurements in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Hala A. Abo el ela, professor, Study Director — faculty of dentistry- Ain shams university
Locations (1):
- faculty of dentistry -Ain shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication